CLINICAL TRIAL: NCT07033832
Title: Acceptance and Commitment Therapy-based Intervention to Decrease Psychological Symptoms and Increase Psychological Flexibility for Parents of a Child With Medical Complexity: a Pilot Randomization-controlled Trial.
Brief Title: Acceptance and Commitment Therapy-based Intervention for Parents of a Child With Medical Complexity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Winsome Lam, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PilotACT
Record Dates: First submitted 2025-06-06; First posted 2025-06-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Acceptance and Commitment Therapy; Child With Medical Complexity; Psychological Flexibility; Randomised Controlled Trial; Depression, Anxiety; Parental Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: single-blinded, pilot randomized controlled trial with two-armed repeated measures
Who Masked: Outcomes Assessor
Masking Description: The project assistant who does not involve in intervention assignment and randomization, will help to conduct the data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-based intervention (Experimental): The ACT-based intervention consists of four face-to-face weekly sessions. Parents in this group will receive two-hour weekly session with the question-and-answer session at the end.
  Interventions: Behavioral: ACT-based intervention
- Control group (No Intervention): Parents of CMC have option to join the usual community social or health care available in the community.

INTERVENTIONS:
Behavioral: ACT-based intervention — Parents in this group will receive two-hour weekly session with the question-and-answer session at the end. The contents of each session are as follows: (1) the first session consist of introductions of ACT, discussion on stress and struggles, and setting homework, (2) the second section includes role play, and the meaning of "value", (3) the third session involves introducing mindfulness of the breath exercise, debrief and homework on practicing mindfulness and (4) the last session includes introduction of "thoughts", and putting values into feasible actions.
  Arms: ACT-based intervention

SUMMARY:
A pilot randomized controlled trial of an Acceptance and Commitment Therapy-based intervention will be conducted to decrease psychological symptoms, while increase psychological flexibility for parents of a child with medical complexity during their difficulties.

DETAILED DESCRIPTION:
Being a parent of the child with medical complexity poses enormous stress because CMC have a chronic complex health condition, which may result in premature death of the CMC. Psychological symptoms commonly experienced by the parents of a CMC. Having a CMC is an ongoing stressor including diagnosis, daily nursing care and symptom management, uncertainty of prognosis that can adequately fear the possibility of relapse. Therefore, seeking an intervention consisting of "Psychological flexibility" is crucial for these parents to manage their stress and difficult emotions more effectively. The ACT intervention help individuals concentrate more on their problems with positive attitude and take initiatives and workable actions to fix the problems associated from the caregiving activities. As a result, they will experience less stress when encountering difficulties and challenges and adapt more effectively. These individuals probably have the potential of natural recoveries from adverse events once the stressor is terminated.

Knowledge gap: A review of the literature reveals a paucity of studies on ACT for Chinese parents of the CMC to decrease their psychological symptoms while enhancing their psychological flexibility in local communities. To fill the knowledge gap, this proposal therefore endeavors to develop an ACT and test its preliminary effects and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* parent of a child with medical complexity aged 1-18
* able to communicate in Chinese and read Chinese
* willing to participate in face-to-face activities

Exclusion Criteria:

* a reported mental health disorder
* engaging in other psychosocial educational programs related to stress reduction
* inability to communicate in Cantonese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The Depression Anxiety Stress Scale (Chinese version) | baseline, week 4
  The DASS is a self-report instrument consisting of 21 items. It is rated on a 4-point scale from 1 (does not apply to me at all) to 4 (applies to me all the time). A higher score on the scale indicates more psychological symptoms.
Psychological flexibility (Chinese version) | baseline, week 4
  The Acceptance and Action Questionnaire-II was used to assess the psychological flexibility of parents. It consists of 7 items and is reported by the parent. Each item is rated on a 7-point Likert scale, ranging from 1 (never true) to 7 (always true).

CONTACTS AND LOCATIONS:
Overall Officials: Winsome LAM, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, China
- School of Nursing The Hong Kong polytechnic university, Kowloon, Hong Kong